CLINICAL TRIAL: NCT02623933
Title: MRI Assisted Focal Boost Integrated With HDR Monotherapy Study in Low and Intermediate Risk Prostate Cancer Patients (MARS)
Brief Title: MRI Assisted Focal Boost With HDR Monotherapy for Prostate Cancer Patients
Acronym: MARS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Andrew Loblaw, Dr Andrew Loblaw, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 222-2015
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: HDR monotherapy; MRI guidance; Intraprostatic lesion; dose paining
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI assisted HDR monotherapy (Experimental): HDR monotherapy to the whole prostate gland (19Gy/1) with MRI assisted focal boost to intraprostatic nodule up to 22.5Gy
  Interventions: Radiation: MRI assisted focal boost with HDR monotherapy

INTERVENTIONS:
Radiation: MRI assisted focal boost with HDR monotherapy — Prior to brachytherapy treatment, a multiparametric MRI will be obtained for identification of the dominant intraprostatic lesion (DIL) and fused with the preplanning transrectal ultrasound. A total of 19 Gy will be prescribed to the prostate, organ at risk limits will be observed and up to 22.5 Gy can be delivered to the DIL

SUMMARY:
Radiation therapy plays an important role in the management of prostate cancer. In recent years it has become evident that higher doses of radiation are required to optimize disease control. The limiting factor of escalating dose to the prostate is the surrounding normal tissue. Despite advances in escalating radiation therapy, failures still occur in 20-30% of patients most often at the site of the original primary disease. As such there is growing interest in further dose escalating to the area of primary disease burden.The aim of this work is to look at the feasibility and toxicities of an integrated focal boost to whole gland prostate treatment using high dose rate brachytherapy.

DETAILED DESCRIPTION:
This study is a pilot study of 60 patients look at the toxicities, biochemical and patient reported quality of life outcomes of an MR-integrated focal boost using HDR prostate brachytherapy. Eligible patients for this study will be determined by pre-brachytherapy MRI (DCE, T2 weighted and diffusion weighted) imaging, to identify a dominant intraprostatic lesion. The HDR dose prescription is 19 Gy to the whole gland ad 22.5 Gy to MRI visible lesion delivered in one fraction, assuming that dose constraints to critical organs can be met.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate
2. Low and Intermediate risk disease defined as T1-T2c, Gleason < 7 and PSA < 20 ng/ml.
3. Prostate volume < 60 cc as determined by US, CT or MRI
4. Ability to undergo MR imaging
5. Provide written informed consent
6. Identified MR nodule (PIRADs 4/5)

Exclusion Criteria:

1. Ineligible for MR imaging due to contraindications
2. Documented nodal or distant metastases
3. Previous pelvic radiotherapy
4. Previous trans-urethral resection of prostate, previous prostatectomy or HIFU
5. Use of androgen deprivation therapy. Use of 5-alpha-reductase inhibitors permitted
6. Poor baseline urinary function defined as International Prostate Symptom Score (IPSS) >15
7. Contra-indication to radical prostate radiotherapy e.g. connective tissue disease or inflammatory bowel disease
8. Significant medical co-morbidity rendering patient unsuitable for general anaesthetic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2027-05-13 (Estimated)

PRIMARY OUTCOMES:
Acute GU and GI toxicities | 3mo
  Measured according to NCI CTCAE v4.0

SECONDARY OUTCOMES:
Late GU and GI toxicities | 5 years
  Measured according to NCI CTCAE v4.0
Quality of life changes | 5 years
  Patient reported outcome utilizing Expanded Prostate Index Composite (EPIC)
Changes in urinary symptoms | 5 years
  Patient reported outcome utilizing International Prostate Symptom Score (IPSS)
Changes in serum prostate-specific antigen (PSA) | 5 years
PSA failure and disease-free survival rates | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided